CLINICAL TRIAL: NCT06120374
Title: Safety and Efficacy of Adjuvant Radioimmunotherapy Compared With Adjuvant Chemotherapy for Upper Tract Urothelial Carcinoma: An Ambispective Cohort Study
Brief Title: Adjuvant Radioimmunotherapy Compared With Adjuvant Chemotherapy for UTUC
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xuesong Li, Department of Urology, Peking University First Hospital
Other Study IDs: LUXUS2.0
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Urothelial Carcinoma
Keywords: upper tract urothelial carcinoma; adjuvant therapy; adjuvant radiotherapy; adjuvant chemotherapy; immunotherapy; safety analysis; progression free survival; overall survival
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Radiotherapy; Drug Therapy; Gemcitabine; Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adjuvant radioimmunotherapy: Participants underwent adjuvant radioimmunotherapy
  Interventions: Radiation: Radiotherapy; Drug: Immunotherapy
- Adjuvant chemotherapy: Participants underwent radical total nephroureterectomy and adjuvant chemotherapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Radiation: Radiotherapy — For participants eligible for enrollment, radiotherapy was started within 4-6 weeks after surgery. Rotational intensity-modulated radiotherapy (VMAT) with daily image-guided radiotherapy (Daily IGRT) technique was used.
  Range of irradiation (patients were randomized into two groups - expanded field irradiation group and involved field irradiation group)
  Other Names: SBRT
  Groups: Adjuvant radioimmunotherapy
Drug: Chemotherapy — For patients eligible for enrollment, postoperative adjuvant chemotherapy was initiated at about 4-6 weeks after surgery, for a total of 4 cycles, with the chemotherapy regimen of gemcitabine + cisplatin. Administration: Gemcitabine 1,000 mg/m2 on days 1 and 8 (completed within 30-60 minutes), cisplatin 70 mg/m2 on day 1.
  Other Names: Based on platinum and gemcitabine
  Groups: Adjuvant chemotherapy
Drug: Immunotherapy — For patients eligible for enrollment, sequential adjuvant immuotherapy was initiated at about 4-6 weeks after surgery, Immunotherapeutic agents include (PD-1/PD-L1) to be used every 21 days postoperatively for one year.
  Other Names: Mainly on PD-1/PD-L1
  Groups: Adjuvant radioimmunotherapy

SUMMARY:
This study is an ambispective cohort observational study to analyze the efficacy of adjuvant radioimmunotherapy (radiotherapy and immunotherapy) compared with adjuvant chemotherapy in patients with the upper urinary tract urothelial carcinoma with high-risk factors (postoperative pathology suggestive of pT2 and above, N+, G3/high-grade and multiple tumors, positive cut margins). A subgroup analysis was performed to obtain the population of patients who might benefit from different treatment approaches. Patients with high risk factors for postoperative recurrence or metastasis will be treated with relevant adjuvant therapy, which in turn will benefit patients.

DETAILED DESCRIPTION:
This study is an ambispective cohort observational study to analyze the efficacy of adjuvant radioimmunotherapy (radiotherapy and immunotherapy) compared with adjuvant chemotherapy in patients with the upper urinary tract urothelial carcinoma with high-risk factors (postoperative pathology suggestive of pT2 and above, N+, G3/high-grade and multiple tumors, positive cut margins). A subgroup analysis was performed to obtain the population of patients who might benefit from different treatment approaches. Patients with high risk factors for postoperative recurrence or metastasis will be treated with relevant adjuvant therapy, which in turn will benefit patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathologic diagnosis as upper urinary tract urothelial carcinoma(UTUC);
* High-risk UTUC: >= pT2, pN+, tumor G3 grade, multifocality or positive surgical margins (according to AJCC 8th edition);
* Aged >= 18 years old;

Exclusion Criteria:

* With Distant metastases already found at the time of surgery; non-R0 resected ;
* History of pelvic and abdominal radiotherapy; history of inflammatory bowel disease; history of systemic chemotherapy;
* Pregnant or lactating women; or women of childbearing potential who are not using reliable contraception;
* History of malignant tumors (except skin cancer that is not malignant melanoma and in situ cervical cancer, tumors that have been cured for more than 5 years);
* Weight loss > 10% within 6 months;
* Existing or coexisting bleeding disorders, active infection;
* Terrible condition cannot tolerate the intervention;
* Unable to sign informed consent due to psychological, family, social and other factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk UTUC patients (met at least one of indications such as: 1. pT2+, 2.G3/High-grade, 3.Multifocality, 4. Positive surgical margin, 5. Positive lymph-node metastasis
Sampling Method: Non-Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-06-08 (Estimated); Study Completion 2029-06-08 (Estimated)

PRIMARY OUTCOMES:
PFS | 1-year, 3-year and 5-year
  Progression-free Survival

SECONDARY OUTCOMES:
OS | 1-year, 3-year and 5-year
  Overall survival
CSS | 1-year, 3-year and 5-year
  Cancer specific survival
LRFS | 1-year, 3-year and 5-year
  Local recurrence free survival
MFS | 1-year, 3-year and 5-year
  Metastasis free survival
IRFS and CRFS | 1-year, 3-year and 5-year
  intravesical-recurrence free survival and contralateral-recurrence free survival

OTHER OUTCOMES:
AE | Peri-therapeutic period
  Adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, M.D., Principal Investigator — Department of Radiotherapy Oncology, Peking University First Hospital; Liqun Zhou, M.D., Study Chair — Department of Urology, Peking University First Hospital
Locations (3):
- China (3):
  - Departmeng of Urology, Peking University First Hospital, Beijing
  - Department of Medical Oncology, Peking University First Hospital, Beijing
  - Department of Radiotherapy Oncology, Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask the prime investigator for the IPD.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within six months after the project completion.
Access Criteria: Not commercial.
URL: http://www.medresman.org.cn/uc/index.aspx

REFERENCES:
- [Background] Seisen T, Krasnow RE, Bellmunt J, Roupret M, Leow JJ, Lipsitz SR, Vetterlein MW, Preston MA, Hanna N, Kibel AS, Sun M, Choueiri TK, Trinh QD, Chang SL. Effectiveness of Adjuvant Chemotherapy After Radical Nephroureterectomy for Locally Advanced and/or Positive Regional Lymph Node Upper Tract Urothelial Carcinoma. J Clin Oncol. 2017 Mar 10;35(8):852-860. doi: 10.1200/JCO.2016.69.4141. Epub 2017 Jan 3. PMID 28045620
- [Background] Birtle A, Johnson M, Chester J, Jones R, Dolling D, Bryan RT, Harris C, Winterbottom A, Blacker A, Catto JWF, Chakraborti P, Donovan JL, Elliott PA, French A, Jagdev S, Jenkins B, Keeley FX Jr, Kockelbergh R, Powles T, Wagstaff J, Wilson C, Todd R, Lewis R, Hall E. Adjuvant chemotherapy in upper tract urothelial carcinoma (the POUT trial): a phase 3, open-label, randomised controlled trial. Lancet. 2020 Apr 18;395(10232):1268-1277. doi: 10.1016/S0140-6736(20)30415-3. Epub 2020 Mar 5. PMID 32145825
- [Result] Li X, Li H, Gao XS, Fang D, Qin S, Zhang Z, Zhou L, Li X, Wang D. Effectiveness of adjuvant radiotherapy for high recurrence risk patients with upper tract urothelial carcinoma. Urol Oncol. 2022 Sep;40(9):410.e1-410.e10. doi: 10.1016/j.urolonc.2022.03.006. Epub 2022 Apr 14. PMID 35431134
- [Result] Li X, Cui M, Gu X, Fang D, Li H, Qin S, Yang K, Zhu T, Li X, Zhou L, Gao XS, Wang D. Pattern and risk factors of local recurrence after nephroureterectomy for upper tract urothelial carcinoma. World J Surg Oncol. 2020 May 30;18(1):114. doi: 10.1186/s12957-020-01877-w. PMID 32473636